CLINICAL TRIAL: NCT01682356
Title: Dietary Nitrate for Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BRJ_201111134
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Hypertension, Pulmonary
Keywords: heart failure; hypertension, pulmonary; oxygen consumption; exercise tolerance
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beetroot juice without nitrate (Placebo Comparator): Patients will be studied before and after ingestion of beetroot juice without nitrate
  Interventions: Dietary Supplement: Beetroot juice
- Beetroot juice with nitrate (Active Comparator): Patients will be studied before and after ingestion of beetroot juice with nitrate.
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — double-blind placebo-controlled cross-over study
  Other Names: Beet It

SUMMARY:
The purpose of this study is to determine if nitrates in a food, in this case - beetroot juice (BRJ) - is efficacious in improving exercise tolerance and/or peak power in patients with heart failure. The investigators will also determine if BRJ improves blood pressure, exercise efficiency, vascular and muscle function, and whether blood levels of nitrates increase hourly for a total of 4 hours after BRJ ingestion. A secondary aim is to determine if BRJ-derived nitrates are still effective at 1, 2 and 4 weeks after starting treatment. A tertiary aim is to determine the variation in the 6 minute walk test. Subjects will answer a basic medical information sheet and undergo a 6-minute walk test. After at least a 48 hours rest, subjects will be asked to repeat the 6 minutes' walk. The investigators will (1) determine if BRJ (as compared to placebo) improves peak power output in heart failure patients and controls (at ~ 1½ to 2 hours after ingestion); (2) compare the changes in cardiac muscle (on average ~ 8-12 hours after) BRJ or placebo ingestion in patients who will be undergoing an left ventricle (LV) assist device placement for clinical purposes. (a cross-sectional study); (3) determine if BRJ decreases elevated pulmonary artery (PA) pressures or improves vascular and/or microvascular function (at ~ 1½ - 2 hours after ingestion) in patients who are already coming in for a PA catheter placement for clinical purposes; (4) compare the physiological changes after BRJ ingestion in non-heart failure control subjects with those of patients with heart failure. Endpoints measured at the same time points after ingestion. The investigators hypothesize (1) that patients with heart failure and controls will have improved exercise capacity and power at lower oxygen cost (and thereby greater efficiency) ~ 1½- 2 hours after ingesting beet juice (BRJ) than after ingesting placebo (beet juice without nitrates); (2) that patients with heart failure will have a greater physiologic response to BRJ than non-heart failure controls since the former have worse physiological function to start with; (3) that patients with high pulmonary artery pressures will have an improvement in the pressures after ingestion with BRJ; (4) that myocardial perfusion will be higher after BRJ ingestion than after placebo; (5) that cyclic guanosine monophosphate (cGMP) levels will be increased in left ventricle assist device (LVAD) samples after BRJ ingestion compared with placebo.

DETAILED DESCRIPTION:
For all studies and sub-studies:

A) All Subjects will be consented. B) All Subjects will give permission for the investigators to review their medical records.

For the BRJ main study (acute dose BRJ intervention):

1. After consenting to participate, subjects will be instructed to refrain from spitting or the use of an antibacterial mouthwash, antacids, proton pump inhibitors, or chewing gum during the study.
2. Subjects will be asked to answer questionnaires regarding their medical health (basic health questionnaire, Minnesota living with heart failure questionnaire, a magnetic resonance safety -i.e., questions regarding implanted pacemakers, etc...) 2a)Subjects will undergo a physical examination at one time during the study.
3. Subjects will be interviewed by a dietician with regards to their typical dietary intake and instructed on a low nitrate diet.
4. In study visit #1 subjects will be randomized to receive either a "shot" of BRJ (James White Drinks)or placebo (BRJ without nitrates).
5. Before and at 3 time points (~hourly) after receiving the BRJ or placebo, subjects will undergo phlebotomy for plasma nutrient/hormone levels and will have their blood pressure checked. They will also be asked to swish (5 minutes) and spit out a dilute ~ 4tbps solution of nitrate,so we can quantify nitrate to nitrite conversion at ~ 1 1/4 hours after ingestion 5A) Subjects will undergo an echocardiogram just after the swish and spit.
6. ~ 1 3/4 hours after ingestion, subjects will undergo a 6 minute walk.
7. ~ 2 hours after ingestion, subjects will pedal an ergometer for 6 min at 15, 30, and 45 W (requiring ~50, ~60, and ~70% of oxygen consumption (VO2) peak, i.e., peak oxygen consumption) while VO2 is measured using a ParvoMedics TrueOne (this is the brand) metabolic cart. Five min of rest will be allowed between stages. The average VO2 during the last 2 min of each stage will be used to calculate gross and delta efficiency using stoichiometric equations as previously described. Following a 10 min rest period, peak power and VO2 peak will determined during a continuous exercise test performed using a 10 W/min ramp protocol.
8. Subjects will then (immediately afterwards )undergo an Magnetic resonance (MR) study of skeletal muscle (and if there is time cardiac performance) with mild exercise (pushing one foot on a pedal for 6 min of submaximal isometric exercise (1 s contraction at 50% of previously-determined maximal voluntary contraction - according to their VO2 peak levels in their medical charts - every 9 s) with spectra acquired before, during, and after exercise.

   During exercise, subjects will have their heart rate, blood pressure and rhythm monitored.
9. Subjects will be asked to undergo a mouth swab for bacterial DNA analyses (after the swish and spit) 9A) Subjects will undergo a Dual-energy Xray absorptiometry (DXA) scan for body composition analysis (either before or after BRJ ingestion - it is a phenotyping measure - not an endpoint)
10. Subjects will undergo a 7 d wash-out period
11. Subjects will come in for study day 2 in which they will receive whichever treatment (BRJ or placebo) that they did not receive at first and then repeat the studies listed above 5)-9).

(The total time of the study is estimated to take 5 hours)

For the longer 2 (or 4) week BRJ substudy: (subjects include HF (heart failure) patients and nonHF controls, i.e., those without heart failure)

1. Subjects will be asked to undergo steps 1-9 above, ingest 1 week of BRJ (1 "shot"/day) and then undergo the studies listed 5)-9).
2. Subjects will be asked to ingest 1 more week of BRJ (1 "shot"/day for a total of 2 weeks) and then undergo a repeat of studies listed 5)-9)

For the BRJ neuromuscular function testing sub-study:

1. Subjects will be asked to undergo steps 1-6 above
2. Subjects will be asked to undergo a mouth swab for bacterial DNA analyses.
3. Subjects will undergo a test of neuromuscular function using an isokinetic dynamometer (a device that measures voluntary muscle force production while controlling the speed of movement) immediately after the echocardiogram at ~2 h after BRJ (or placebo ingestion).

3A) Subjects will be asked to undergo an optional skeletal muscle biopsy immediately after the Biodex study.

3B) Subjects will undergo a dual-energy isokinetic dynamometry study for body composition analysis (at any time point during the study day).

4) Subjects will undergo a 7 d washout period.

5) Subjects will come in for Study day 2 in which they will receive whichever treatment (BRJ or placebo) they did not receive at first and then repeat the studies listed above 1-3.

For the Pulmonary artery (PA) pressure sub-study:

NOTE: This study will only be performed in patients who are undergoing a PA catheter placement for clinical purposes (high PA pressures) anyway.

1. After consenting to participate, subjects will be instructed to refrain from spitting or the use of an antibacterial mouthwash, antacids, proton pump inhibitors, or chewing gum during the study.
2. Subjects will be asked to answer questionnaires regarding their medical health (basic health questionnaire, Minnesota living with heart failure questionnaire, etc.) 2a) Subjects will be asked to undergo a physical examination.
3. Before and at 3 (hourly) time points after receiving a "shot" of BRJ, subjects will undergo phlebotomy for plasma nutrient/hormone levels and will have their blood pressure checked and will blow into a tube connected to a small machine that will measure the amount of nitric oxide in their breath. Subjects will also have cardiovascular measurements (e.g., cardiac output, PA pressure, etc.) made before and at 3 ~ hourly time points after receiving the BRJ. These measurements will be made using a PA catheter that is being placed for clinical purposes.
4. If a subject is to undergo an LVAD placement he/she will be randomized to receive BRJ or placebo the evening before surgery (anticipated average ~ 8-12 hours before), and then the LV core will be harvested and immediately frozen for later analysis.
5. Subjects who will be undergoing myocardial perfusion studies will undergo the same basic studies (breath NO, plasma nitrate/nitrite determination, as mentioned in the neuromuscular aim, but subjects will also undergo a positron emission tomography (PET) study in which they will receive O-15 water for quantification of myocardial blood flow ~ 2 hours after consumption of BRJ or placebo. Then they will undergo a washout phase of 7 d and then repeat the PET study after the other treatment (BRJ or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Men and women will have a history of heart failure (and/or pulmonary hypertension for PA catheter substudy).
* Age > or = 18 y and controls of the same age range without heart failure.

Exclusion Criteria:

* Age < 18 y.
* Those taking phosphodiesterase inhibitors (e.g., Viagra) will be excluded, as these can potentiate NO effects.
* Those taking proton pump inhibitors, antacids, or xanthine oxidase inhibitors will be excluded as these can affect reduction of nitrate (NO3-) and nitrite (NO2-) to nitric oxide (NO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Peterson, MD, Principal Investigator — Washington University School of Medicine; Andrew R Coggan, PhD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Purdue University Indianapolis, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No
Aggregate data that contains no HIPPA identifiers will be made available as required if the request complies with all federal and University policies for data sharing. IPD will not be shared since this is a small study at a single institution, so the likelihood of identifying subjects would be increased.

REFERENCES:
- [Background] Masschelein E, Van Thienen R, Wang X, Van Schepdael A, Thomis M, Hespel P. Dietary nitrate improves muscle but not cerebral oxygenation status during exercise in hypoxia. J Appl Physiol (1985). 2012 Sep 1;113(5):736-45. doi: 10.1152/japplphysiol.01253.2011. Epub 2012 Jul 5. PMID 22773768
- [Background] Hobbs DA, Kaffa N, George TW, Methven L, Lovegrove JA. Blood pressure-lowering effects of beetroot juice and novel beetroot-enriched bread products in normotensive male subjects. Br J Nutr. 2012 Dec 14;108(11):2066-74. doi: 10.1017/S0007114512000190. Epub 2012 Mar 14. PMID 22414688
- [Background] Cermak NM, Gibala MJ, van Loon LJ. Nitrate supplementation's improvement of 10-km time-trial performance in trained cyclists. Int J Sport Nutr Exerc Metab. 2012 Feb;22(1):64-71. doi: 10.1123/ijsnem.22.1.64. PMID 22248502
- [Background] Vanhatalo A, Fulford J, Bailey SJ, Blackwell JR, Winyard PG, Jones AM. Dietary nitrate reduces muscle metabolic perturbation and improves exercise tolerance in hypoxia. J Physiol. 2011 Nov 15;589(Pt 22):5517-28. doi: 10.1113/jphysiol.2011.216341. Epub 2011 Sep 12. PMID 21911616
- [Background] Kenjale AA, Ham KL, Stabler T, Robbins JL, Johnson JL, Vanbruggen M, Privette G, Yim E, Kraus WE, Allen JD. Dietary nitrate supplementation enhances exercise performance in peripheral arterial disease. J Appl Physiol (1985). 2011 Jun;110(6):1582-91. doi: 10.1152/japplphysiol.00071.2011. Epub 2011 Mar 31. PMID 21454745
- [Background] Ferreira LF, Behnke BJ. A toast to health and performance! Beetroot juice lowers blood pressure and the O2 cost of exercise. J Appl Physiol (1985). 2011 Mar;110(3):585-6. doi: 10.1152/japplphysiol.01457.2010. Epub 2010 Dec 23. No abstract available. PMID 21183624
- [Background] Vanhatalo A, Bailey SJ, Blackwell JR, DiMenna FJ, Pavey TG, Wilkerson DP, Benjamin N, Winyard PG, Jones AM. Acute and chronic effects of dietary nitrate supplementation on blood pressure and the physiological responses to moderate-intensity and incremental exercise. Am J Physiol Regul Integr Comp Physiol. 2010 Oct;299(4):R1121-31. doi: 10.1152/ajpregu.00206.2010. Epub 2010 Aug 11. PMID 20702806
- [Background] Wilkerson DP, Hayward GM, Bailey SJ, Vanhatalo A, Blackwell JR, Jones AM. Influence of acute dietary nitrate supplementation on 50 mile time trial performance in well-trained cyclists. Eur J Appl Physiol. 2012 Dec;112(12):4127-34. doi: 10.1007/s00421-012-2397-6. Epub 2012 Apr 20. PMID 22526247
- [Background] Bailey SJ, Winyard P, Vanhatalo A, Blackwell JR, Dimenna FJ, Wilkerson DP, Tarr J, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of low-intensity exercise and enhances tolerance to high-intensity exercise in humans. J Appl Physiol (1985). 2009 Oct;107(4):1144-55. doi: 10.1152/japplphysiol.00722.2009. Epub 2009 Aug 6. PMID 19661447
- [Derived] Tawa M, Nagata R, Sumi Y, Nakagawa K, Sawano T, Ohkita M, Matsumura Y. Preventive effects of nitrate-rich beetroot juice supplementation on monocrotaline-induced pulmonary hypertension in rats. PLoS One. 2021 Apr 8;16(4):e0249816. doi: 10.1371/journal.pone.0249816. eCollection 2021. PMID 33831045
- [Derived] Coggan AR, Leibowitz JL, Spearie CA, Kadkhodayan A, Thomas DP, Ramamurthy S, Mahmood K, Park S, Waller S, Farmer M, Peterson LR. Acute Dietary Nitrate Intake Improves Muscle Contractile Function in Patients With Heart Failure: A Double-Blind, Placebo-Controlled, Randomized Trial. Circ Heart Fail. 2015 Sep;8(5):914-20. doi: 10.1161/CIRCHEARTFAILURE.115.002141. Epub 2015 Jul 15. PMID 26179185

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Nitrate: Acute (single dose) placebo, 7 day washout, acute (single dose) nitrate
- Nitrate Then Placebo: Acute (single dose) nitrate, 7 day washout, acute (single dose) placebo
Period: Overall Study
Arm/Group | Placebo Then Nitrate | Nitrate Then Placebo
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Nitrate: Placebo then nitrate
- Nitrate Then Placebo: Nitrate then placebo
- Total: Total of all reporting groups
Arm/Group | Placebo Then Nitrate | Nitrate Then Placebo | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12) | 57 (12) | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximal Knee Extensor Power
Description: Maximal power of the quadriceps muscle group as measured using isokinetic dynamometry
Time Frame: 2-3 h after acute dose of beetroot juice containing or essentially devoid of nitrate
Population: Only 9 participants were assessed for maximal knee extensor power.
Measure: Mean (Standard Error); unit: W/kg
Groups:
- Placebo: Beetroot juice without nitrate.
- Nitrate: Beetroot juice with nitrate.
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 9 | 9
W/kg | 4.20 (0.33) | 4.74 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.0153, t-test, 2 sided; Paired

2. Secondary Outcome: VO2peak
Description: Peak oxygen consumption as measured during semi-recumbent cycle ergometer exercise
Time Frame: 2-3 h after acute dose of beetroot juice containing or essentially devoid of nitrate
Population: Only 8 participants were assessed for VO2peak.
Measure: Mean (Standard Error); unit: mL/min/kg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 8 | 8
mL/min/kg | 21.4 (2.1) | 23.0 (2.3)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.0131, t-test, 2 sided; Paired

3. Other Pre Specified Outcome: Baseline Plasma Nitrate
Description: Nitrate in plasma before ingestion of beetroot juice
Time Frame: 0 h
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
umol/L | 27 (4) | 31 (4)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.83, ANOVA — P value adjusted for multiplicity; Plasma nitrate values were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

4. Other Pre Specified Outcome: Plasma Nitrate @ 1 h
Description: Nitrate in plasma 1 h after ingestion of beetroot juice
Time Frame: 1 h
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
umol/L | 25 (3) | 334 (31)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p < 0.0000001, ANOVA — P values adjusted for multiplicity. Exact P value 6.06 x 10^-18; Plasma nitrate values were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

5. Other Pre Specified Outcome: Plasma Nitrate @ 2 h
Description: Nitrate in plasma 2 h after ingestion of beetroot juice
Time Frame: 2 h
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
umol/L | 24 (3) | 386 (172)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p < 0.0000001, ANOVA — P values adjusted for multiplicity. Exact P value 1.87 x 10^-20; Plasma nitrate values were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

6. Other Pre Specified Outcome: Plasma Nitrate @ 10 Min Post-exercise
Description: Nitric oxide in breath 10 min after completion of exercise testing
Time Frame: 10 min post-exercise
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
umol/L | 25 (3) | 397 (45)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p < 0.0000001, ANOVA — P values adjusted for multiplicity. Exact P value 8.23 x 10^-21; Plasma nitrate values were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

7. Other Pre Specified Outcome: Baseline Plasma Nitrite
Description: Nitrite in plasma before ingestion of beetroot juice
Time Frame: 0 h
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
umol/L | 0.292 (0.070) | 0.341 (0.146)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.6847, ANOVA — P values adjusted for multiplicity; Plasma nitrate values were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

8. Other Pre Specified Outcome: Plasma Nitrite @ 1 h
Description: Nitrite in plasma 1 h after ingestion of beetroot juice
Time Frame: 1 h
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
umol/L | 0.254 (0.064) | 0.298 (0.085)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.6847, ANOVA — P values adjusted for multiplicity; Plasma nitrate values were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

9. Other Pre Specified Outcome: Plasma Nitrite @ 2 h
Description: Nitrite in plasma 1 h after ingestion of beetroot juice
Time Frame: 2 h
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
umol/L | 0.216 (0.050) | 0.315 (0.059)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.4078, ANOVA — P values adjusted for multiplicity; Plasma nitrate values were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

10. Other Pre Specified Outcome: Plasma Nitrite @ 10 Min Post-exercise
Description: Nitrite in plasma 10 min after completion of exercise testing
Time Frame: 10 min post-exercise
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
umol/L | 0.306 (0.083) | 0.400 (0.093)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.4078, ANOVA — P values adjusted for multiplicity; Plasma nitrate values were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

11. Other Pre Specified Outcome: Baseline Breath Nitric Oxide
Description: Nitric oxide in breath before ingestion of beetroot juice
Time Frame: 0 h
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 15 | 15
ppm | 18 (1) | 20 (2)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.3042, ANOVA — P value adjusted for multiplicity; Breath nitric oxide values were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

12. Other Pre Specified Outcome: Breath Nitric Oxide @ 1 h
Description: Nitric oxide in breath 1 h after ingestion of beetroot juice
Time Frame: 1 h
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 15
ppm | 19 (2) | 29 (3)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p < 0.0000001, ANOVA — P value adjusted for multiplicity. Exact P value 3.469 x 10^-7; [statistical method as in outcome 11, analysis 1]

13. Other Pre Specified Outcome: Breath Nitric Oxide @ 2 h
Description: Nitric oxide in breath 2 h after ingestion of beetroot juice
Time Frame: 2 h
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 15
ppm | 19 (2) | 31 (3)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p < 0.0000001, ANOVA — P value adjusted for multiplicity. Exact P value 7.202 x 10^-8; [statistical method as in outcome 11, analysis 1]

14. Other Pre Specified Outcome: Breath Nitric Oxide @ 10 Min Post-exercise
Description: Nitric oxide in breath 10 min after completion of exercise testing
Time Frame: 10 min post
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 15
ppm | 17 (1) | 27 (3)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.00000213, ANOVA — P value adjusted for multiplicity. Exact P value 2.129 x 10^-6; [statistical method as in outcome 11, analysis 1]

15. Other Pre Specified Outcome: Baseline Systolic Blood Pressure
Description: Systolic blood pressure before ingestion of beetroot juice
Time Frame: 0 h
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
mmHg | 106 (4) | 109 (4)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.3918, ANOVA — P values adjusted for multiplicity; Values for blood pressure were analyzed using a repeated measures ANOVA followed by Holm-Šídák multiple comparison testing

16. Other Pre Specified Outcome: Systolic Blood Pressure @ 1 h
Description: Systolic blood pressure 1 h after ingestion of beetroot juice
Time Frame: 1 h
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
mmHg | 104 (4) | 109 (3)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.05980, ANOVA — P values adjusted for multiplicity; [statistical method as in outcome 15, analysis 1]

17. Other Pre Specified Outcome: Systolic Blood Pressure @ 2 h
Description: Systolic blood pressure 2 h after ingestion of beetroot juice
Time Frame: 2 h
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
mmHg | 104 (3) | 106 (4)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.3918, ANOVA — P values adjusted for multiplicity; [statistical method as in outcome 15, analysis 1]

18. Other Pre Specified Outcome: Systolic Blood Pressure @ 10 Min Post-exercise
Description: Systolic blood pressure 10 min after completion of exercise testing
Time Frame: 10 min post-exercise
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
mmHg | 111 (4) | 106 (3)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.09870, ANOVA — P values adjusted for multiplicity; [statistical method as in outcome 15, analysis 1]

19. Other Pre Specified Outcome: Baseline Diastolic Blood Pressure
Description: Diastolic blood pressure before ingestion of beetroot juice
Time Frame: 0 h
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
mmHg | 68 (3) | 71 (3)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.6044, ANOVA — P values adjusted for multiplicity; [statistical method as in outcome 15, analysis 1]

20. Other Pre Specified Outcome: Diastolic Blood Pressure @ 1 h
Description: Diastolic blood pressure 1 h after ingestion of beetroot juice
Time Frame: 1 h
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
mmHg | 66 (3) | 68 (2)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.6044, ANOVA — P values adjusted for multiplicity; [statistical method as in outcome 15, analysis 1]

21. Other Pre Specified Outcome: Diastolic Blood Pressure @ 2 h
Description: Diastolic blood pressure 2 h after ingestion of beetroot juice
Time Frame: 2 h
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
mmHg | 67 (3) | 68 (2)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.8819, ANOVA — P values adjusted for multiplicity; [statistical method as in outcome 15, analysis 1]

22. Other Pre Specified Outcome: Diastolic Blood Pressure @ 10 Min Post-exercise
Description: Diastolic blood pressure 10 min after completion of exercise testing
Time Frame: 10 min post-exercise
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nitrate
Number analyzed (Participants) | 17 | 17
mmHg | 69 (3) | 69 (2)
Statistical Analysis 1: Comparison: Placebo vs Nitrate; Test type: Superiority; p = 0.8987, ANOVA — P values adjusted for multiplicity; [statistical method as in outcome 15, analysis 1]

23. Other Pre Specified Outcome: Cardiac Function
Description: Subjects undergoing MRI or echocardiography will have various measures of cardiac function made
Time Frame: after ingestion of BRJ or placebo
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Pulmonary Artery Pressure
Description: Each patient who is going to have a PA catheter placed for clinical purposes will have their PA pressures measured before and after ingestion of BRJ.
Time Frame: 1 day intervention
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Vascular Function
Description: Each subject undergoes a laser Doppler test and a brachial artery test after ingesting BRJ or placebo. There is a 10 d washout period and then the test is repeated after the subject ingests the BRJ or placebo (whichever was not taken the first time).
Time Frame: each patient will undergo a study for a maximum of ~ 2 weeks
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Myocardial Perfusion
Description: We will measure perfusion using noninvasive PET imaging
Time Frame: before and after BRJ or placebo ingestion
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Myocardial Tissue Changes
Description: We will measure cyclic GMP and nitrate in LV tissue after LVAD placement and after ingestion of either BRJ or placebo
Time Frame: after BRJ or placebo ingestion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: One day per intervention with 7 days of washout in between
Description: Adverse event reporting used definitions from clinicaltrials.gov
Arm/Group | Placebo | Nitrate
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Due to restrictions on research resulting from the COVID-19 pandemic, many outcome measures/planned substudies were not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT01682356/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT01682356/SAP_001.pdf